CLINICAL TRIAL: NCT02914899
Title: Informing the Adaptation of a CHW Model to Facilitate Lung Cancer Screening for the Chinese Community
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-949
Record Dates: First submitted 2016-09-21; First posted 2016-09-26 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer Screening; Current or Past Cigarette Smoker
Keywords: Professional Drivers; 16-949
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

ARMS (5):
- Pilot RCT Control Group (Active Comparator): Eligible NYC Chinese livery drivers will receive written materials only
  Interventions: Behavioral: Surveys
- Pilot RCT CHW Intervention Group (Experimental): Eligible NYC Chinese livery drivers will receive written materials and navigation for shared decision making (SDM) and lung cancer screening (LCS).
  Interventions: Behavioral: Surveys; Behavioral: Navigation
- Focus Group (Experimental): The investigators conducted a series of 4-6 focus groups with Chinese livery drivers who (currently, or in the past) smoke.
  Interventions: Behavioral: Focus groups
- In-Depth Interview Group (Experimental): 12-15 in-depth interviews with livery base management and staff, and with 12-15 primary care physicians (PCPs), clinic directors, hospital CFOs, heads of financial services and counseling, and heads of radiology facilities serving the Chinese community.
  Interventions: Behavioral: In-depth interviews
- Pre-pilot Group (Experimental): Approximately 10 Chinese livery drivers who smoke or who quit smoking with the past 15 years and have a 30 pack-year history of smoking
  Interventions: Behavioral: Surveys; Behavioral: Navigation

INTERVENTIONS:
Behavioral: Surveys — Intake surveys recorded demographics, workplace profile, financial profile, health care access, cancer screening behavior, medical history, etc.
  Exit surveys asked whether drivers received shared decision making (SDM) counseling, completed LCS (low-dose computed tomography [LDCT] scan), had barriers, felt satisfied, etc.
  Arms: Pilot RCT CHW Intervention Group; Pilot RCT Control Group; Pre-pilot Group
Behavioral: Navigation — CHWs facilitated SDM and LCS for drivers, providing navigation ( finding a PCP, scheduling appointments, assisting with insurance, etc.), following up on results and next steps.
  Arms: Pilot RCT CHW Intervention Group; Pre-pilot Group
Behavioral: Focus groups — Gained drivers' perspectives on adapting the community health worker (CHW) model to facilitate lung cancer screening (LCS).
  Arms: Focus Group
Behavioral: In-depth interviews — Interviews with Chinese livery bases elicited perspectives on adapting the CWH model for the drivers' occupational environment.
  Interviews with PCPs, clinic directors, etc. serving Chinese communities provided insight into adapting the CHW model within the health care context.
  Arms: In-Depth Interview Group

SUMMARY:
The purpose of this study is to test if our Community Health Worker program can help at-risk NYC Chinese community members participate in shared decision making and lung cancer screening (if appropriate) and compare it to the help provided by written materials.

DETAILED DESCRIPTION:
The study first used qualitative methods to inform the adaptation of a CHW model to facilitate lung cancer screening completion in an extremely high-risk group, NYC Chinese livery drivers who smoke or who quit within the past 15 years. A series of focus groups with Chinese livery drivers who smoke, a series of in-depth interviews with livery base management and staff, primary care physicians (PCPs), clinic directors, hospital CFOs, heads of financial services and counseling, and heads of radiology facilities serving the Chinese community were conducted to explore barriers and factors related to cancer screening. Findings were used to develop adapted intervention materials, including a CHW Manual for Facilitating Shared Decision Making and Lung Cancer Screening. Once adaptation is complete, the researchers will conduct a pre-pilot to refine the adapted CHW intervention materials. The researchers will then conduct a pilot randomized controlled trial (RCT) to assess the feasibility of the refined CHW model (intervention) versus written materials (control) to facilitate SDM and LCS (when appropriate) in an extremely high-risk group, NYC Chinese livery drivers eligible (by USPTSF criteria) for LCS. Feasibility results will be used to inform the planning and design of large scale RCTs, targeting Chinese drivers, as well as other driver populations in NYC and throughout the U.S., and other high risk Chinese smoking populations in other occupations (e.g. restaurant work, construction). The study is currently in the pre-pilot phase and expects to launch the pilot phase by the summer of 2020. Due to the effects of the COVID-19 crisis, the researchers have extended the pre-pilot participation time frame to 12 months. The study population has also indicated concern to attend doctor's appointments for SDM/LCS during COVID-19. As such, MSK is extending the study time frame to an additional 6 months. . CHWs will also be hosting health education workshops at community organizations, family associations, and public libraries. These workshops will be conducted in English, Mandarin, and Cantonese and cover topics including smoking cessation and lung cancer screening.

ELIGIBILITY:
Inclusion Criteria:

Focus Group Participants:

* Of Chinese descent
* Non-U.S. born
* Fluent in Mandarin
* Livery driver
* Age 45-80
* Current or past (within 15 years) cigarette smoker (no specific pack year requirement)

In Depth Interview Participants Livery Staff

* Of Chinese descent
* Non-U.S. born
* Fluent in Mandarin
* Livery base owner or employee
* Age ≥ 21

Health Care Providers and Administrators:

* Primary care physician, clinic director, hospital administrator, or radiology facility or department administrator
* Age ≥ 21
* Fluent in English

CHW pre-pilot RCT participants:

* Of Chinese descent
* Fluent in Mandarin
* Male
* Livery driver
* Age 55-80 years old
* Driven for 3 months or longer
* 30 pack year history
* Current smoker or quit within 15 years
* Will not be traveling out of New York Area for more than 1 month in the next 3 months

CHW pilot RCT participants

* Of Chinese descent
* Fluent in Mandarin or Cantonese
* Male
* Professional driver
* Age 50-80 years old
* Driven for 3 months or longer
* Last drove professionally within the last 18 months with plans of returning
* 20 pack year smoking history
* Current smoker or quit within 15 years
* Will not be traveling out of New York Area for more than 3 months in the next 12 months
* Has not completed LDCT in the past year.

Exclusion Criteria:

* Has a household member who has already participated (or agreed to participate).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
(Pre-Pilot Phase) Increased uptake in SDM and LCS | 2 years
  To determine whether participation in the interventions leads to increased completion of SDM and LCS with LDCT.
(Pilot Phase) Increased uptake in SDM and LCS | 2 years
  To determine whether participation in the interventions leads to increased completion of SDM and LCS with LDCT.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Leng, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT02914899/ICF_000.pdf